CLINICAL TRIAL: NCT02216188
Title: Phase IB Follow-up, Randomized, Controlled, Parallel Group, Patient-blinded, Single-center Study to Assess One Boost With AFFITOPE® PD01A With Regard to Safety/Tolerability, Immunological + Clinical Activity in Patients Who Have Received the Vaccine Within the Study AFF008
Brief Title: Follow-up Study to Assess One Boost Immunization With AFFITOPE® PD01A With Regard to Safety and Clinical Activity
Acronym: AFF008A
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Affiris AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AFFiRiS 008A; 2014-002489-54 (EudraCT Number)
Record Dates: First submitted 2014-08-12; First posted 2014-08-13 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A: AFFITOPE® PD01A + Adjuvant (Experimental): one injection of 15µg AFFITOPE® PD01A/ adjuvanted
  Interventions: Biological: AFFITOPE® PD01A
- B: AFFITOPE® PD01A + Adjuvant (Experimental): one injection of 75µg AFFITOPE® PD01A/ adjuvanted
  Interventions: Biological: AFFITOPE® PD01A
- Control (Other): Untreated control group
  Interventions: Other: Control

INTERVENTIONS:
Biological: AFFITOPE® PD01A — s.c. injection
  Arms: A: AFFITOPE® PD01A + Adjuvant; B: AFFITOPE® PD01A + Adjuvant
Other: Control — Untreated control group
  Arms: Control

SUMMARY:
This is a follow-up study to assess safety and clinical activity of continued AFFITOPE® PD01A vaccinations in patients with Parkinson's disease. Patients, who have already participated in AFF008 will be involved and will be receive one boost immunization with AFFITOPE® PD01A. One study site in Vienna (Austria) will be involved.

In addition, up to 8 patients will be offered participation within an untreated control group.

ELIGIBILITY:
Inclusion Criteria:

* Prior participation in AFF008 and AFF008E
* Written informed consent signed and dated by the patient and the caregiver (caregiver is not mandatory)
* In the investigator's opinion, does not have visual or auditory impairments that would reduce the patients' ability to complete study questionnaires or be unable to receive instructions for these
* Female patients of childbearing potential are eligible if they use a medically accepted contraceptive method
* Stable doses of PD medications for at least 3 months prior to Visit 0 and during the entire trial period and of all other medications for at least 30 days prior to Visit 1 if considered relevant by the investigator

Exclusion Criteria:

* Women of childbearing potential without birth control or pregnant women
* Participation in another clinical trial (except AFF008E) within 3 months before Visit 0
* History of questionable compliance to visit schedule; patients not expected to complete the clinical trial
* Autoimmune disease or allergy to components of the vaccine
* History of cancer (Exceptions: basal cell carcinoma, intraepithelial cervical neoplasia)
* Active infectious disease
* Immunodeficiency
* Significant systemic illness or psychiatric illness
* Alcoholism or substance abuse
* Prior treatment with experimental immunotherapeutics for PD including IVIG (with the exception of AFFITOPE ® PD01A), with immunosuppressive drugs or treatment with deep brain stimulation
* Venous status rendering it impossible to place an i.v. access

Ages: 40 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-08; Primary Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Tolerability | 6 month
  * Occurrence of any Adverse Events (AE)
  * Occurrence of any Serious Adverse Events (SAE)
  * Withdrawal criteria (number of patients who withdraw due to AEs/ reason for withdrawal)

SECONDARY OUTCOMES:
Immunological | 6 month
  - Titer of antibodies specific for the immunizing peptide, KLH (keyhole limpet hemocyanin; carrier protein), aSynuclein (aSyn), bSyn, aggregated aSyn as assessed by ELlSA, FACS (or equivalent methods)

OTHER OUTCOMES:
Clinical Activity | 6 month
  * Change in motor symptoms (MDS-UPDRS III)
  * Change in non-motor PD symptoms (e.g.; MDS-UPDRS Ia, II, PDQ39, PD NMS, cognition)
  * Change in biological and radiological markers (e.g. CSF alpha synuclein Levels in cerebrospinal fluid)

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Volc, Prim, Dr., Principal Investigator — Studienzentrum der PROSENEX, AmbulatoriumbetriebsgesmbH an der Confraternität-Privatklinik Josefstadt, Skodagasse 32, 1080 Vienna
Locations (1):
- Studienzentrum der PROSENEX, AmbulatoriumbetriebsgesmbH an der Confraternität-Privatklinik Josefstadt, Skodagasse 32, 1080 Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Derived] McFarthing K, Simuni T. Clinical Trial Highlights: Targetting Alpha-Synuclein. J Parkinsons Dis. 2019;9(1):5-16. doi: 10.3233/JPD-189004. No abstract available. PMID 30741694